CLINICAL TRIAL: NCT07289672
Title: Förändrat Livsmedelsval Vid Inflammatorisk Tarmsjukdom
Brief Title: Food Limitations In Crohn's Disease and Ulcerative coliTis
Acronym: FLIT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-04814-01
Record Dates: First submitted 2025-11-19; First posted 2025-12-17 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-10

CONDITIONS: Crohn Disease (CD); Ulcerative Colitis (UC); IBD (Inflammatory Bowel Disease)
Keywords: IBD; ulcerative colitis; Crohn's disease; nutritional intervention
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Diet; Educational Status

STUDY DESIGN:
Who Masked: Participant
Masking Description: Although the patients know that they will be given dietary advice they will not know what type of intervention the other group will be offered. Since dietary advice must be given by the investigators the study cannot be blinded to them.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normal diet (No Intervention)
- Test diet calprotectin (Experimental)
  Interventions: Other: Diet
- Test diets Nordic (Experimental)
  Interventions: Other: Diet
- Digital information tool (Experimental)
  Interventions: Other: education

INTERVENTIONS:
Other: Diet — Healthy nordic based food
  Arms: Test diet calprotectin; Test diets Nordic
Other: education — Digital information tool/education on food in inflammatory bowel disease (IBD)
  Arms: Digital information tool

SUMMARY:
The goal of this clinical trial is to increase the knowledge on what type of diet affects inflammation and how to better convay that information in patients with inflammatory bowel disease (IBD) and decrease selective eating in patients with IBD. The main questions it aims to answer are:

* will the use of calprotectin as a control for changes in inflammation decrease selective food choices?
* will the use of a digital information tool increase quality of life (QoL) och decrease selctive eating patterns?
* will a diet based on nordic food choices decrease inflammation and increase QoL?

Researchers will compare with IBD-patients in ordinary care.

Participants will eat a test diet during six weeks or go through a digital information tool.

DETAILED DESCRIPTION:
Patients with inflammatory bowel disease attending the out-patient clinic at Skåne university hospital with calprotectin 200-600 will be invited to participate in this diet intervention study. They will be divided into four arms with 35 patients in each, normal diet, test diets or diet with digital information tool.

The diet will be recorded at study start and end with a food diary for four days, as will health related quality of life. The patients clinical characteristics (demographics) and disease activity (diarrhoea frequency, blood in stools, abdominal pain, CRP and calprotectin) will be recorded.

The patients clinical characteristics (demographics) and disease activity (diarrhoea frequency, blood in stools, abdominal pain, CRP and calprotectin) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Ulcerative colitis and Crohn's disease
* Calprotectin 200-600

Exclusion Criteria:

* Non-active disease
* solely procitis
* Severe disease
* past extensive bowel surgery
* treatment with antibiotics (last month or present)
* pregnancy
* unability to understand spoken or written Swedish
* Multimorbidity which aggrevate participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Concentration of calproteictin | From enrollment until 6 weeks

SECONDARY OUTCOMES:
Four days registrered food intake | At beginning and after 6 week
  Food intake will be registrered at beginning and after 6 week

CONTACTS AND LOCATIONS:
Locations (1):
- Mag- och tarmmottagningen, Skåne university hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No